CLINICAL TRIAL: NCT02923375
Title: An Open-Label Phase 1 Study to Investigate the Safety and Efficacy of CYP-001 for the Treatment of Adults With Steroid-Resistant Acute Graft Versus Host Disease
Brief Title: A Study of CYP-001 for the Treatment of Steroid-Resistant Acute Graft Versus Host Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cynata Therapeutics Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CYP-GvHD-P1-01; 2016-000070-38 (EudraCT Number)
Record Dates: First submitted 2016-10-03; First posted 2016-10-04 (Estimated); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Graft vs Host Disease
MeSH Terms: conditions — Graft vs Host Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Cohort A (Experimental): Mesenchymoangioblast-derived mesenchymal stem cells (CYP-001) at a dose of 1 million cells/kg (up to a maximum of 100 million cells) by IV infusion on two occasions (Day 0 and Day 7)
  Interventions: Biological: Mesenchymoangioblast-derived mesenchymal stem cells
- Cohort B (Experimental): Mesenchymoangioblast-derived mesenchymal stem cells (CYP-001) at a dose of 2 million cells/kg (up to a maximum of 200 million cells) by IV infusion on two occasions (Day 0 and Day 7)
  Interventions: Biological: Mesenchymoangioblast-derived mesenchymal stem cells

INTERVENTIONS:
Biological: Mesenchymoangioblast-derived mesenchymal stem cells — The active agent in CYP-001 is allogeneic mesenchymoangioblast-derived mesenchymal stem cells (MCA-derived MSCs), which are produced using the proprietary Cymerus™ platform technology. Cymerus™ refers to the process of generating cell-based products from intermediate cells, MCAs, which in turn are derived from induced pluripotent stem cells or iPSCs. The iPSCs used in the Cymerus™ process were derived from blood donated by a fully-consented healthy adult donor, and were reprogrammed using a transgene-free, viral-free and feeder-free technique.
  Other Names: CYP-001

SUMMARY:
The purpose of this study is to assess the safety, tolerability and efficacy of two infusions of CYP-001 in adults with steroid-resistant GvHD.

DETAILED DESCRIPTION:
This is a multi-centre, open label, dose escalation study to assess the safety, tolerability and efficacy of two infusions of CYP-001, in adults who have steroid-resistant GvHD.

Participants will receive standard of care treatment throughout the study, according to local procedures. The first eight participants will be enrolled in Cohort A and receive a CYP-001 dose of 1 million cells per kg, up to a maximum dose of 100 million cells, on Day 0 and Day 7. Subject to a safety review of data from Cohort A, an additional eight participants will be enrolled into Cohort B and receive a CYP-001 dose of 2 million cells/kg, up to a maximum dose of 200 million cells, on Day 0 and Day 7. The primary evaluation period concludes for each participant 100 days after the first dose of CYP-001. Participants will have study visits on Days 0, 3, 7, 14, 21, 28, 60 and 100. Subsequently, participants will enter a long term follow-up period, which concludes 2 years after the first dose of CYP-001.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis using consensus grading with steroid-resistant Grade II-IV acute GvHD, after a haematopoietic stem cell transplant for a haematological disorder.
* Life expectancy of at least one month.
* Agree to have follow-up data collected for two years after their initial dose of CYP-001 (under a separate protocol).

Exclusion Criteria:

* Pregnant or breastfeeding or plan to become pregnant within three months of receiving their last dose of CYP-001.
* Have received any investigational research agent within 30 days or five half-lives (whichever is longer) prior to the first dose of IMP.
* Known or suspected current alcohol or substance abuse problem.
* Progressive or relapsing haematological malignancy, a current solid tumour, or previous malignant solid tumour that is likely to recur during the period of the study (with the exception of a past history of basal or squamous cell carcinomas).
* Heart failure (NYHA Functional Class II-IV) and/or pulmonary failure.
* Haemodynamically unstable and/or at high risk of cardiovascular events.
* Terminal organ failure.
* Meningitis, pneumonia with hypoxemia, HIV or another severe or uncontrolled systemic infection, which in the opinion of the investigator is likely to impact on the ability of the patient to participate in the trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-08-28 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of treatment emergent adverse events [safety and tolerability] | 28 days
  Safety
Incidence and severity of serious adverse events deemed possibly related to CYP-001 [safety and tolerability] | 100 days
  Safety

SECONDARY OUTCOMES:
Complete Response by Day 28 | 28 days
  Proportion of participants who show a Complete Response (absence of any signs or symptoms of GvHD) by Day 28
Partial Response by Day 28 | 28 days
  Proportion of participants who show a Partial Response (improvement in the severity of GvHD by at least one grade compared to baseline) by Day 28
Overall Survival at Day 28 | 28 days
  Proportion of participants who survive until Day 28
Complete Response by Day 100 | 100 days
  Proportion of participants who show a Complete Response by Day 100
Partial Response by Day 100 | 100 days
  Proportion of participants who show a Partial Response by Day 100
Overall Survival at Day 100 | 100 days
  Proportion of participants who survive until Day 100

CONTACTS AND LOCATIONS:
Overall Officials: Kilian Kelly, PhD, Study Director — Cynata Therapeutics Limited
Locations (7):
- Australia (2):
  - Sydney Local Health District, Sydney, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
- United Kingdom (5):
  - NHS Foundation Trust, Bristol
  - NHS Trust, Leeds
  - NHS Foundation Trust, Liverpool
  - NHS Foundation Trust, Manchester
  - NHS Foundation Trust, Nottingham

REFERENCES:
- [Derived] Kelly K, Bloor AJC, Griffin JE, Radia R, Yeung DT, Rasko JEJ. Two-year safety outcomes of iPS cell-derived mesenchymal stromal cells in acute steroid-resistant graft-versus-host disease. Nat Med. 2024 Jun;30(6):1556-1558. doi: 10.1038/s41591-024-02990-z. Epub 2024 May 22. PMID 38778211
- [Derived] Bloor AJC, Patel A, Griffin JE, Gilleece MH, Radia R, Yeung DT, Drier D, Larson LS, Uenishi GI, Hei D, Kelly K, Slukvin I, Rasko JEJ. Production, safety and efficacy of iPSC-derived mesenchymal stromal cells in acute steroid-resistant graft versus host disease: a phase I, multicenter, open-label, dose-escalation study. Nat Med. 2020 Nov;26(11):1720-1725. doi: 10.1038/s41591-020-1050-x. Epub 2020 Sep 14. PMID 32929265